CLINICAL TRIAL: NCT04196972
Title: Transforming Professional Engagement, Practice Efficiency, and Community Building Through Team Meetings in a Telementoring Environment
Brief Title: Telementoring Intervention (ECHO) for the Transformation of Professional Engagement, Practice Efficiency, and Community Building Through Team Meetings in Diagnostic Imaging Clinicians
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0639; NCI-2019-07565 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0639 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-12-02; First posted 2019-12-12 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (ECHO telementoring) (Experimental): Participants attend ECHO telementoring sessions over 1 hour weekly for 13 weeks.
  Interventions: Other: Communication Intervention; Other: Questionnaire Administration
- Arm B (wait-list, ECHO telementoring) (Experimental): Participants are placed on a wait-list for 13 weeks and then attend ECHO telementoring sessions over 1 hour weekly for 13 weeks.
  Interventions: Other: Communication Intervention; Other: Questionnaire Administration; Other: Waiting List

INTERVENTIONS:
Other: Communication Intervention — Receive ECHO telementoring intervention
Other: Questionnaire Administration — Ancillary studies
Other: Waiting List — Placed on wait-list
  Other Names: Waitlist
  Arms: Arm B (wait-list, ECHO telementoring)

SUMMARY:
This trial studies how well the Extension for Community Healthcare Outcomes (ECHO) telementoring intervention works in transforming professional engagement, practice efficiency, and community building through team meetings in diagnostic imaging clinicians. This study may help researchers learn more about the potential benefits of a model for team meetings aimed at bringing physicians together from multiple practice locations when few opportunities exist for meaningful, collegial interactions. It may also help diagnostic imaging clinicians engage more effectively with colleagues at distant sites and become more engaged with their work.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of the proposed anti-burnout intervention for faculty at MD Anderson, defined as at least 35/50 of participants each attending at least 9 out of 13 sessions.

SECONDARY OBJECTIVES:

I. To explore any changes in burnout, measured by the Maslach Burnout Inventory (MBI) and Mini-Z surveys.

II. To explore any changes in the self-reported health status of participants, as measured by the RAND Short-Form 36 (SF36) survey.

III. To understand participants' perception of the benefits and usefulness of the intervention, measured by the customized Globalized Perception/Impression of Benefits Survey.

IV. To define methods for improving the intervention, based on participants' feedback following each session.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM A: Participants attend ECHO telementoring sessions over 1 hour weekly for 13 weeks.

ARM B: Participants are placed on a wait-list for 13 weeks and then attend ECHO telementoring sessions over 1 hour weekly for 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Faculty must be diagnostic imaging clinicians with a primary appointment in the Division of Diagnostic Imaging at MD Anderson

Exclusion Criteria:

* Faculty that have an official leadership role (Division Head or Department Chair)
* Faculty that have previously participated in any previous live ECHO clinic or ECHO activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of sessions attended | through study completion, an average of 1 year
  Will be evaluated by attendance records for each session. Will estimate the attendance rate (p = proportion of participants attending at least 9 out of 13 sessions) with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org